CLINICAL TRIAL: NCT02712619
Title: An Open-label, Parallel Group Clinical Trial to Investigate the Pharmacokinetics/Pharmacodynamics of 250/1000 mg of Metformin IR After Oral Administration in Healthy Male Volunteers
Brief Title: Pharmacokinetic-Pharmacodynamic Relationship of Metformin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, MD, PhD, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP0
Record Dates: First submitted 2016-02-22; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

ARMS (2):
- metformin 250mg (Experimental): metformin 375/250 mg
  Interventions: Drug: Metformin
- metformin 1000mg (Experimental): metformin 1000/1000 mg
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Two doses of metformin with 12 hour interval

* low dose group (375/250 mg)
* high dose group (1000/1000mg)

DETAILED DESCRIPTION:
A study to evaluate and compare the pharmacokinetic-pharmacodynamic relationship between different metformin dose groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 45
* Body weight 50 to 100 kg
* fasting serum glucose 70 to 125 mg/dL
* who provide informed consent voluntarily

Exclusion Criteria:

* any significant renal, gastrointestinal, hepatic, and metabolic condition
* any co/prior medication within 14 days of study drug administration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration | 0-12 hour
Area under the metformin concentration curve | 0-12 hour
Area under the glucose curve | 2-5 hour

REFERENCES:
- [Derived] Chung H, Oh J, Yoon SH, Yu KS, Cho JY, Chung JY. A non-linear pharmacokinetic-pharmacodynamic relationship of metformin in healthy volunteers: An open-label, parallel group, randomized clinical study. PLoS One. 2018 Jan 17;13(1):e0191258. doi: 10.1371/journal.pone.0191258. eCollection 2018. PMID 29342199